CLINICAL TRIAL: NCT04494724
Title: A Phase 2 Trial to Evaluate the Safety and Tolerability of Clazakizumab® [Anti-Interleukin (IL)-6 Monoclonal] Compared to Placebo for the Treatment of COVID-19 Infection
Brief Title: Clazakizumab vs. Placebo - COVID-19 Infection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00025969
Record Dates: First submitted 2020-07-21; First posted 2020-07-31 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: COVID-19 Infection
Keywords: COVID-19; coronavirus infection; respiration, artificial; extracorporeal membrane oxygenation; randomized controlled trial; respiratory distress syndrome, adult
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Respiratory Aspiration; Respiratory Distress Syndrome | interventions — clazakizumab

STUDY DESIGN:
Intervention Model Description: This single-site, phase 2 randomized, double-blind, placebo-controlled trial is designed to administer a single dose of clazakizumab or placebo on day 0. If, after 24 hours or up to 14 days from the first infusion, the participant's condition worsens or does not improve, the investigator may elect to provide a single, open-label dose of clazakizumab regardless of the initial group assignment. All except the investigational pharmacist will remain blinded as to the initial group assignment until data lock.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinded to all except investigational pharmacy. Only the optional second infusion, if determined necessary to administer, will be open-label. The patient and study team will remain blinded until data lock at the end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Clazakizumab (Experimental): Clazakizumab - 25mg in 50 milliliters (mL) of 0.9% saline, IV infusion over 30 minutes.
  Interventions: Drug: Clazakizumab
- Placebo (Placebo Comparator): Placebo - 50 mL 0.9% saline, IV infusion over 30 minutes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clazakizumab — Infusion
  Arms: Clazakizumab
Drug: Placebo — Infusion
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effectiveness and safety of treatment with clazakizumab compared to a placebo (inactive substance). We are proposing to try this drug to treat coronavirus disease 2019 (COVID-19) infection. Patients with COVID-19 infection have been shown to have increases in certain inflammatory processes. Clazakizumab is an antibody (immune system protein) that blocks certain inflammatory processes. The treatment plan is to attempt to inhibit or block these inflammatory processes in order to try to limit the damage COVID-19 causes to the lungs.

DETAILED DESCRIPTION:
The purpose of this randomized, double-blind, placebo-controlled trial is to evaluate the safety and efficacy of clazakizumab vs placebo for the prevention of acute respiratory distress syndrome (ARDS) in patients with COVID-19 and pulmonary manifestations. The study will compare clazakizumab to placebo in a randomized, double-blind fashion followed by an open-label dose of clazakizumab if there is no improvement or a worsening of condition occurs after 24-hours or anytime during the first 14 days after the first dose of clazakizumab or placebo. We hypothesize that clazakizumab will be safely tolerated and will reduce the risk of progression of COVID-19 to acute respiratory distress syndrome.

Primary Objective:

• To evaluate the safety and tolerability of clazakizumab vs placebo for the treatment of patients with COVID-19 disease and signs of pulmonary involvement

Sixty adult patients with COVID-19 and signs of pulmonary involvement at Houston Methodist who are not in need of ventilator support at the time of enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 at the time of screening.
2. Participant or legally authorized representative (LAR) must be able to understand and provide informed consent.
3. Hospitalized with coronavirus disease (COVID-19) confirmed by polymerase chain reaction (PCR) assay from any specimen (eg, respiratory, blood, urine, stool, other bodily fluid) within the prior 72 hours.
4. C-reactive protein (CRP) > 3.5 mg/dL
5. Evidence of pulmonary involvement with at least 2 of the following:

   1. oxygen saturation at rest in ambient air with peripheral capillary oxygen saturation (SpO2) ≤ 94%
   2. tachypnea with resting respiration rate > 25 breaths/minute
   3. Partial pressure of oxygen (PaO2)/initial fraction of inspired oxygen (FiO2) ≤ 300 mmHg
   4. Chest imaging (radiograph, CT, or ultrasound) with abnormalities consistent COVID-19 pneumonia

Exclusion Criteria:

1. Previous hypersensitivity or allergic reactions to clazakizumab
2. Lactating or pregnant females
3. Patients with latent tuberculosis (TB) and who are not receiving treatment
4. Patients with active TB
5. Patients with known active inflammatory bowel disease, untreated diverticulitis, or gastrointestinal perforation
6. Requiring mechanical ventilation or extracorporeal membrane oxygenation (ECMO)
7. A significantly abnormal general serum screening lab result defined as a white blood cell (WBC) count < 3.0 X 10^3/mL, a hemoglobin (Hgb) < 8.0 g/dL, a platelet count < 50 X 10^3/mL, an aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 5 times upper limit normal
8. Participation in another clinical trial investigating COVID-19-aimed agents
9. Presence of any medical or psychosocial condition, which the investigator believes, would hinder adherence to the study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-07-13 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | 24 hours
  Proportion of participants who experience treatment-related adverse events (TEAE) ≥ Grade 3 (CTCAE v5.0) during the first 24 hours after infusion of clazakizumab or placebo

SECONDARY OUTCOMES:
Requirement for mechanical ventilation and/or extracorporeal membrane oxygenation (ECMO) | 14 days
  Proportion of participants who need mechanical ventilation and/or extracorporeal membrane oxygenation (ECMO) after the first dose of clazakizumab or placebo
Infusion-related reactions during 24 hours from the time of infusion | 24 hours
  Proportion of participants who experience infusion-related reactions during the first 24 hours after infusion of clazakizumab or placebo
Patient survival at 28 days | 28 days
  Proportion of participants alive at day 28 after the first dose of clazakizumab or placebo
Patient survival at 60 days | 60 days
  Proportion of participants alive at day 60 after the first dose of clazakizumab or placebo
Requirement for open-label clazakizumab | 14 days
  Proportion of participants who require an open-label dose of clazakizumab
Time in the intensive care unit (ICU) | 60 days
  Number of days in the ICU following the first dose of clazakizumab or placebo
Time in the hospital | 60 days
  Number of days in the hospital following the first dose of clazakizumab or placebo
Time to mechanical ventilation | 60 days
  Number of days from first dose of clazakizumab or placebo to requiring mechanical ventilation
Clinical status improvement assessed by the World Health Organization (WHO) Clinical Progression Scale at day 14 | 14 days
  Difference in WHO Clinical Progression Scale between clazakizumab and placebo
Clinical status improvement assessed by World Health Organization (WHO) Clinical Progression Scale at day 28 | 28 days
  Difference in WHO Clinical Progression Scale between clazakizumab and placebo
Change in Radiologic Assessment of Lung Edema (RALE) at day 14 | 14 days
  Difference in mean or median change in radiologic assessment of lung edema (RALE) score at day 14 from baseline between clazakizumab or placebo
Change in Radiologic Assessment of Lung Edema (RALE) at day 28 | 28 days
  Difference in mean or median change in radiologic assessment of lung edema (RALE) score at day 28 from baseline between clazakizumab or placebo

CONTACTS AND LOCATIONS:
Overall Officials: Howard Huang, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jones SA, Jenkins BJ. Recent insights into targeting the IL-6 cytokine family in inflammatory diseases and cancer. Nat Rev Immunol. 2018 Dec;18(12):773-789. doi: 10.1038/s41577-018-0066-7. PMID 30254251
- [Result] Tanaka T, Kishimoto T. Targeting interleukin-6: all the way to treat autoimmune and inflammatory diseases. Int J Biol Sci. 2012;8(9):1227-36. doi: 10.7150/ijbs.4666. Epub 2012 Oct 24. PMID 23136551
- [Result] Uciechowski P, Dempke WCM. Interleukin-6: A Masterplayer in the Cytokine Network. Oncology. 2020;98(3):131-137. doi: 10.1159/000505099. Epub 2020 Jan 20. PMID 31958792
- [Result] Ruan Q, Yang K, Wang W, Jiang L, Song J. Correction to: Clinical predictors of mortality due to COVID-19 based on an analysis of data of 150 patients from Wuhan, China. Intensive Care Med. 2020 Jun;46(6):1294-1297. doi: 10.1007/s00134-020-06028-z. PMID 32253449
- [Result] Gao Y, Li T, Han M, Li X, Wu D, Xu Y, Zhu Y, Liu Y, Wang X, Wang L. Diagnostic utility of clinical laboratory data determinations for patients with the severe COVID-19. J Med Virol. 2020 Jul;92(7):791-796. doi: 10.1002/jmv.25770. Epub 2020 Apr 10. PMID 32181911
- [Result] Le RQ, Li L, Yuan W, Shord SS, Nie L, Habtemariam BA, Przepiorka D, Farrell AT, Pazdur R. FDA Approval Summary: Tocilizumab for Treatment of Chimeric Antigen Receptor T Cell-Induced Severe or Life-Threatening Cytokine Release Syndrome. Oncologist. 2018 Aug;23(8):943-947. doi: 10.1634/theoncologist.2018-0028. Epub 2018 Apr 5. PMID 29622697
- [Result] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Result] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343